CLINICAL TRIAL: NCT06224959
Title: Prevalence of Migraine and Neuropathic Pain in Osteoarthritis: Multicenter, Multidisciplinary, Cross-sectional Epidemiological Study.
Brief Title: Migraine and Neuropathic Pain in Osteoarthritis
Acronym: MEDUSA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2023 MATHIEU; 2023-A00093-42 (Other: ANSM)
Record Dates: First submitted 2024-01-08; First posted 2024-01-25 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis; Migraine; Neuropathic Pain
Keywords: osteoarthritis; migraine; neuropathic pain
MeSH Terms: conditions — Osteoarthritis; Migraine Disorders; Neuralgia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to estimate the frequency of neuropathic pain and migraines in a group of patients with osteoarthritis of the knees, hips, hands, spine or other joints. In addition to their usual care for osteoarthritis, participants will complete questionnaires to define migraine and neuropathic pain.

DETAILED DESCRIPTION:
This study will be proposed to patients with osteoarthritis who come for their routine consultation. If the patient has no abjection to taking part in the study, the doctor will give them the questionnaires to fill in. The questionnaires are about: perception of pain , depression and anxiety, how patients manage their disease emotionally, migraine, neuropathic pain, functional ability, osteoarthritis assessment.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years old
* patients with articular or/and spinal osteoarthritis
* affiliation to a social security system.
* able to read and understand french

Exclusion Criteria:

* patients who refuse to participate in the study
* patients unable to complete self-questionnaires
* minors or adults under the protection of the law or under the protection of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with articular and/or spinal osteoarthritis, under the care of the University Hospital of Clermont-Ferrand (Rheumatology, Physical Medicine and Rehabilitation, Sports Medicine, Occupational Health and Environment, Orthopedics), and/or managed by specialized professionals (general practitioners, sports physicians, rheumatologists, rehabilitation specialists, orthopedic surgeons) in private medical practice
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2028-03-27 (Estimated); Study Completion 2028-03-27 (Estimated)

PRIMARY OUTCOMES:
the presence of neuropathic pain in patients | 10 minutes
  Neuropathic pain is defined by a "Douleur Neuropathique" (DN)-4 questionnaire given to the patients, A patient is considered to have characteristics of neuropathic pain if their DN-4 questionnaire score is greater than 4.
  DN-4 is a questionnaire used to estimate the likelihood of neuropathic pain in patients and to aid in the diagnosis of neuropathic pain. There are 4 items with a total of 10 questions, the patient must answer yes or no to each question and the doctor counts the answers at the end of the questionnaire, 1 for a yes answer and 0 for a no answer, and the sum obtained is the patient's score.
the presence of migraine in patients | 10 minutes
  Completing the headache questionnaire of the International Headache Society (IHS). Strict migraine is defined as meeting all the criteria for migraine as defined by the IHS. Probable migraine sufferers are those who meet all but one of the migraine criteria.
  IHS criteria is defined by :
  A. At least five seizures meeting criteria B through D.
  B. Headache attacks lasting 4 to 72 hours (without treatment).
  C. Headache with at least two of the following features : One-sided; pulsating; moderate or severe; worsened by routine physical activities, such as climbing or descending stairs
  D. At least one of the following during the headache :nausea and/or vomiting; photophobia and phonophobia.
  E. Clinical examination should be normal between attacks. In case of doubt, an organic disorder must be excluded by appropriate additional investigations.

SECONDARY OUTCOMES:
the presence of anxiety and depression symptoms in patients | 10 minutes
  to evaluate the impact of migraine or/and neuropathic pain in patients with osteoarthritis on anxiety and depression symptoms by the Hospital Anxiety and Depression scale questionnaire (HADs). The HADs questionnaire have 14 items, each item is rated on a scale of 0 to 3, with higher scores associated with the presence and level of symptoms.
measure the level of catastrophizing thoughts related to pain in patients | 10 minutes
  to assess how patients with osteoarthritis perceive and react to pain emotionally because of their migraine or/and neuropathic pain by the Pain Catastrophizing Scale (PCS) questionnaire. The questionnaire have 13 items that assess 3 components of catastrophization pain : exaggeration, rumination and helplessness.
Impact of headhache in patients | 10 minutes
  Headache patients complete the Headache Impact Test (HIT-6), which measures the impact of headaches on daily life. It's a 6-question questionnaire with a choice of 5 answers, with points ranging from 6 to 13 per answer. The scores for each column of each question are added together. The higher the score, the greater the impact of the headache on daily life. Scores range from 36 to 78.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain MATHIEU, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France, France